CLINICAL TRIAL: NCT05722821
Title: Effects of Hypopressive Abdominal Gymnastics (GAH) in Spanish Postmenopausal Women With Urinary Incontinence: A Randomized Clinical Trial
Brief Title: Effects of Hypopressive Abdominal Gymnastics in Urinary Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jaén (Other)
Responsible Party: Principal Investigator, Agustín Aibar Almazán, Principal investigator, University of Jaén
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: - University of Jaén.
Record Dates: First submitted 2023-02-01; First posted 2023-02-10 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Menopause; Older Adults

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: For the assignment to the groups, a random sampling will be carried out using the Epidat program. This classification will be hidden, therefore, those responsible for admitting the patients to the intervention phase will not know to which group each one has been assigned. Said assignment will be made previously by a researcher who will not intervene in the subsequent phases of evaluation, data recording intervention and database preparation. The assignment will be communicated using fully opaque sealed envelopes. The analysis of the results will be carried out by a researcher unrelated to the group assignment and the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): An experimental group (GE): that after an initial evaluation will be subjected to a hypopressive abdominal gymnastics program, for 12 weeks with 2 weekly sessions (Tuesday and Thursday, controlling adherence to the sessions through attendance), with a duration of 45 min per session. Once the intervention is finished, you will be subjected to a final evaluation to see if there is a difference or not with the results obtained at the beginning.
  Interventions: Other: Hypopressive intervention
- Control group (No Intervention): A control group (CG): that will not be subjected to treatment, which will be evaluated in the pre and post phase of the study, and a follow-up by telephone contact of adherence to physical activity. The participants assigned to this group will receive general advice on the positive effects of the regular practice of physical activity aimed at preventing urinary incontinence, and they will be given the guide of recommendations for the promotion of physical activity.

INTERVENTIONS:
Other: Hypopressive intervention — Hypopressive abdominal gymnastics is based on a basic level hypopressive exercise program that will be:
  * A duration of 12 weeks with a frequency of 2 sessions a week and lasting 45 minutes each. Hypopressive abdominal exercises will be performed individually adapted to the capacity of the participant.
  * There will be an initial anatomical training of the muscles involved in carrying out the exercise and practice in the respiratory technique for a duration of 15 minutes. Afterwards, hypopressive exercises will begin for 20-30 minutes, changing positions if possible.
  Arms: Experimental group

SUMMARY:
The increase in the age of the population is a problem that affects both Spain and the rest of the world. Life expectancy increases, and this will influence the quality of life that older people will have. The quality of life is related to the health of the population. Women live longer than men and have diseases such as urinary incontinence that are more frequent in them. This is related to childbirth, increasing age, and menopause due to the hormonal level. Therefore, there are a series of problems related to both physical and mental health associated both with increasing age and with the situation of hormonal change that occurs after the onset of menopause. All of this will influence deficient pelvic musculature, sexual function, sleep quality, and depression/anxiety. Conservative treatment using hypopressive abdominal exercises has been shown to be beneficial at the level of health in female populations with urinary incontinence. The challenge lies in designing exercise programs that, in addition to achieving these benefits, are attractive with acceptance and adherence. The objective of this doctoral thesis is to study the effects of hypopressive abdominal exercises for 12 weeks on quality of life related to urinary incontinence in women, sleep quality, anxiety and depression, and female sexual function in women. Spanish postmenopausal women.

DETAILED DESCRIPTION:
Society is facing a longer life expectancy due to improvements in medicine, which leads to an increase in the aging population. According to the National Institute of Statistics (INE), the population over 65 years of age has been increasing from 2001 to 2020, assuming a growth of 14.6% in Europe and 13.6% in Spain. Demographic indicators indicate a greater increase in life expectancy in women (from 82.7-85.1 years) than in men (75.9-79.6 years).

Currently, women present more specific health problems than men due to their physiological conditions, such as the menopausal transition. At the vasomotor level, hot flashes or hot flashes form the most distinctive element of this stage at the sexual level, such as the lack of lubrication, discomfort or pain, and altered function; on a psychological level, anxiety and depression, which is a syndrome linked to disorders such as sadness and its impact on menopause, is quite significant; and the affectation of sleep that are one of the main complaints of women at this stage. All these symptoms affect the quality of life of women both physically and mentally.

With aging and the incidence of menopause, a series of changes in women's health take place, constituting a natural and inevitable process; which can cause unwanted events, such as urinary incontinence. UI is defined as the involuntary loss of urine, within urinary incontinence the most prevalent is stress urinary incontinence (SUI) in 10-30% in most studies, and compared to men 75% of women are more affected than men. This condition can cause disorders in the quality of life, and among the main risk factors are increasing age, parity, family history of prolapse, obesity, lifting heavy objects and constipation also influences. Women with prolapses may present with vaginal, bladder, bowel, back, abdominal, and sexual symptoms. Women frequently suffer from UI due to atrophic changes in the urogenital tract. Therefore, a conservative treatment where the evaluation of the pelvic floor strength and the functional use of pelvic floor muscle training are previously carried out is recommended to achieve health benefits and therefore quality of life.

Recent studies have shown that women with pelvic floor dysfunctions who perform pelvic floor muscle training through hypopressive abdominal exercises improve the pelvic muscles and quality of life of postmenopausal women with UI and prolapses. The hypopressive abdominal exercises (AHT) technique can be classified as a breathing exercise. It was developed by Dr. Marcel Caufriez, a physical therapist in 1980. This inventor theorized that the decrease in abdominal pressure obtained with AHT may produce reflex activation of the abdominal wall and pelvic floor muscles, thus reducing UI and prolapses. The AHT, in summary, involves diaphragmatic breathing, total air breathing, and gradual contraction of the transverse abdominis and intercostal muscles with rise in the diaphragm and apnea. This conservative treatment technique is adaptable to the mind (since you have to concentrate on breathing) and body integration exercise that can be worked on anywhere and anytime, without the need for special equipment.

The directors of this doctoral thesis have experience in this field, with several works published in journals located in the first tercile and quartile of their categories according to the JCR index.

ELIGIBILITY:
Inclusion Criteria:

* Women with urinary incontinence with cessation of menstrual activity for 12 months or more and who are able to understand the instructions and exercise protocols of this project.

Exclusion Criteria:

* Contraindications for physical tests, cancer or serious illness, musculoskeletal and neurological diseases (Parkinson's disease, multiple sclerosis, diabetic neuropathy, cerebrovascular accident, etc.).
* Taking drugs that affect the central nervous system or antidepressants, or lack of willingness to participate in the study.
* People who have previously carried out pelvic floor reeducation programs.

Min Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Gender Based: Yes
Enrollment: 112 (Actual)
Dates: Start 2023-03-13 (Actual); Primary Completion 2023-06-02 (Actual); Study Completion 2023-06-12 (Actual)

PRIMARY OUTCOMES:
International Consulation on Incontinence Short Quality of Life Questionnaire | Up to twelve weeks
  Is a brief questionnaire aimed at measuring the perception of UI symptoms and the patient's quality of life. The scores of the questions 1+2+3 are added.
  Any score greater than zero is considered a diagnosis of UI.
PSQI (Pittsburgh Sleep Quality Index) | Up to twelve weeks
  A simple and valid assessment of both sleep quality and disturbance that might affect. They consist of 10 questions divided into four subscales: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep discomfort, medication use and daytime dysfunctions, adding up to a total score. The higher value represents a worse result. Higher scores indicate poorer sleep.
Pelvic organ prolapse/urinary incontinence sexual function questionnaire-12 | Up to twelve weeks
  It is an instrument with adequate psychometric characteristics to assess sexual function in women with pelvic floor problems in Spain. The score is made by adding the scores of each item, (from 0=always to 4=never), inverting this score for items 1, 2, 3, and 4.
Prolapse quality of life questionnaire | Up to twelve weeks
  The P-QoL questionnaire is a self-reported tool that contains 20 questions representing nine quality of life domains: general health (1 item), prolapse impact (1 item), role limitations (2 items), physical limitations (2 items), social limitations (3 items), personal relationships (2 items), emotions (3 items), sleep/energy (2 items) and severity measures (4 items). Scores in each domain range from 0 to 100. Higher scores indicate a greater impairment of quality of life, and lower scores indicate a good quality of life. Additionally, there are 18 questions regarding urinary, bowel, and prolapse/vaginal symptoms, which do not have an assigned score. Response options are on a Likert scale with ranges between 1 and 4, except for the first question, that ranges between 1 and 5. Symptoms questions and personal relationships domains offer the option Not applicable.
Handgrip Strength | Up to twelve weeks
  Dynamometer will be employed to assess hand grip strength.
TUG test (Timed Up and Go test) | Up to twelve weeks
  Is a simple test used to assess a person's mobility and physical function.
Chair sit and reach test. | Up to twelve weeks
  To test low back and hamstring flexibility.
Back scratch test. | Up to twelve weeks
  To measure general shoulder range of motion.

SECONDARY OUTCOMES:
BMI (Body Mass Index) | Up to twelve weeks
  Is calculated from the formula, Weight (kg) / Height2 (m2), whose unit is kg/m2. It is a rough indicator of total body fat.
Waist circumference. | Up to twelve weeks
  Is used to assess central fat distribution and degree of abdominal obesity.
Hip circumference | Up to twelve weeks
  It is the greatest circumference of hip.
Waist-to-hip ratio. | Up to twelve weeks
  Is the dimensionless ratio of the circumference of the waist to that of the hips. This is calculated as waist measurement divided by hip measurement.

CONTACTS AND LOCATIONS:
Locations (1):
- Center for the Elderly "Gallur", Zaragoza, Spain